CLINICAL TRIAL: NCT02177617
Title: Synergistic Effects of Neurotoxin and Physical Therapy
Brief Title: Neurotoxin and Physical Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: American Academy of Neurology (Other); National Ataxia Foundation (Other); American Brain Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB201400343
Record Dates: First submitted 2014-06-13; First posted 2014-06-27 (Estimated); Results first posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-08

CONDITIONS: Cervical Dystonia
Keywords: Cervical Dystonia; Botox
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A; Neurotoxins; Physical Therapy Modalities; Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Botox only (Active Comparator): Participants randomized to receive Botox injections alone.
  Interventions: Drug: Botox injection; Procedure: Transcranial magnetic stimulation (TMS)
- Botox plus Physical Therapy (Active Comparator): Participants randomized to receive Botox injection combined with Physical Therapy
  Interventions: Drug: Botox injection; Behavioral: Physical Therapy; Procedure: Transcranial magnetic stimulation (TMS)

INTERVENTIONS:
Drug: Botox injection — Participants will receive a tailored dose of Botox to address their Cervical Dystonia symptoms
  Other Names: Neurotoxin
Behavioral: Physical Therapy — Participants will undergo physical therapy sessions with a physical therapist trained in movement disorders. Participants will be instructed to continue these exercises five times per week, and will be called weekly by the investigator to check progress.
  Arms: Botox plus Physical Therapy
Procedure: Transcranial magnetic stimulation (TMS) — For these tests, participants will sit in a chair that looks like one found at the dentist's office. A nerve stimulator will be placed on the wrist of the right hand to stimulate the median and ulnar nerves. The intensity of the nerve stimulator will be gradually increased until the right thumb begins to twitch. A magnetic coil will be placed on the scalp on the left side of the head, overlying the brain's motor cortex, to stimulate the brain's output to the muscles in the opposite hand. This procedure will be repeated using the left wrist and the right side of the head.

SUMMARY:
This study aims to compare Botox injections without Physical Therapy sessions to Botox injections combined with Physical Therapy sessions for treatment of Cervical Dystonia. It is expected that Botox combined with Physical Therapy will improve Cervical Dystonia symptoms and quality of life more than Botox alone. It is also expected that Botox combined with Physical Therapy will enhance neuroplasticity, or the ability of the brain to make new connections, more than Botox alone at 4-5 weeks, and remain improved at 12 weeks, after Botox injection.

DETAILED DESCRIPTION:
The study will recruit primary cervical dystonia patients (age 18-80) who are stable on Allergan botulinum toxin type A (Botox). Patients will be randomized to receive their typical Botox injection alone, or with physical therapy.

At Baseline, disease characteristics (as measured by the Toronto Western Spasmodic Torticollis Rating Scale, or TWSTRS, and the Clinical Global Impression of Severity, or CGIS) will be measured, along with quality of life (from the Short Health 36 Survey Form 36, or SF-36). One subscale of the TWSTRS will be videotaped to be later evaluated by blinded movement disorder specialists. A pain scale will also be completed and range of head motion will be measured using a device similar to a protractor (called a goniometer). An individualized Botox injection will be administered, as well as transcranial magnetic stimulation (TMS) to measure neuroplasticity, or the ability of the brain to make new connections. If randomized to receive physical therapy, participants will also receive instructions to perform physical therapy exercises five times per week by a physical therapist who specializes in movement disorders. The investigator will call weekly to check how the participant is doing with the exercise program.

The same procedures outlined above will also be performed at 5 weeks past baseline, and at 12 weeks (except for the Botox injection, which will only be given at baseline and 12 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-80 with a diagnosis of Cervical Dystonia, which will be confirmed by a movement disorders specialist
* Positive response to at least two prior treatments with Botox as indicated by an improvement in Clinical Global Improvement Scale.
* Received last dose of Botox a minimum of 12 weeks prior to baseline visit.

Exclusion Criteria:

* Any conditions that would contraindicate transcranial magnetic stimulation (for example, pregnancy or epilepsy)
* Any secondary, fixed, post-traumatic, or psychogenic dystonia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12; Primary Completion 2017-01-07 (Actual); Study Completion 2017-01-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aparna Wagle Shukla, MD, Principal Investigator — University of Florida; Michael S Okun, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Botox Only | Botox Plus Physical Therapy
Started | 8 | 8
Completed | 8 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Botox Only | Botox Plus Physical Therapy | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 5 | 5 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.3 (5.2) | 64.7 (5.4) | 64.5 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 4 | 4 | 8
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16
TWSTRS pain [Mean (Standard Deviation); unit: units on a scale] | 4 (1.4) | 3.8 (1.5) | 3.8 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS)
Description: The Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) is a measure of symptoms, pain, and disability related to Cervical Dystonia. The total TWSTRS scale includes a global outcome score (total score) and scores on each of 3 subscales for severity (0-35), disability (0-30), and pain (0-20), which are summed together for a total score (0-85), with higher scores indicating greater impairment. The TWSTRS is completed by a neurologist who visually assesses the patient's symptoms, and asks the patient to self-report on pain and disability.
Time Frame: absolute value at Week 12
Population: mean difference between two groups was calculated
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Botox Only | Botox Plus Physical Therapy
Number analyzed (Participants) | 8 | 8
total score on a scale | 28 (10.2) | 20.1 (9.8)

2. Primary Outcome: SF-36 Physical Functioning Subscore
Description: The Short Form 36-Item Health Scale (SF-36) is a health survey with 36 questions that is self-reported by the study participant. It contains 8 subscales, one of which is Physical Functioning, calculated from 10 of the 36 questions. Different questions have different score ranges and valences. Therefore, their response for each question is linearly transformed to a value of 0-100 (for example, choosing response 3 on a scale of 1-5 is transformed to 60). These ten values are then averaged to generate the Physical Functioning subscore, ranging from 0-100. The higher the response value and the subscore, the higher degree of physical functioning.
  More details on RAND SF-36 scoring here: https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form/scoring.html
Time Frame: absolute value at Week 12
Population: mean difference between two groups calculated
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Botulinum Only: Participants randomized to receive Botulinum injections alone.
  Botulinum injection: Participants will receive a tailored dose of Botulinum to address their Cervical Dystonia symptoms
  Transcranial magnetic stimulation (TMS): For these tests, participants will sit in a chair that looks like one found at the dentist's office. A nerve stimulator will be placed on the wrist of the right hand to stimulate the median and ulnar nerves. The intensity of the nerve stimulator will be gradually increased until the right thumb begins to twitch. A magnetic coil will be placed on the scalp on the left side of the head, overlying the brain's motor cortex, to stimulate the brain's output to the muscles in the opposite hand. This procedure will be repeated using the left wrist and the right side of the head.
- Botulinum Plus Physical Therapy: Participants randomized to receive Botulinum injection combined with Physical Therapy
  Botulinum injection: Participants will receive a tailored dose of Botulinum to address their Cervical Dystonia symptoms
  Physical Therapy: Participants will undergo physical therapy sessions with a physical therapist trained in movement disorders. Participants will be instructed to continue these exercises five times per week, and will be called weekly by the investigator to check progress.
  Transcranial magnetic stimulation (TMS): For these tests, participants will sit in a chair that looks like one found at the dentist's office. A nerve stimulator will be placed on the wrist of the right hand to stimulate the median and ulnar nerves. The intensity of the nerve stimulator will be gradually increased until the right thumb begins to twitch. A magnetic coil will be placed on the scalp on the left side of the head, overlying the brain's motor cortex, to stimulate the brain's output to the muscles in the opposite hand. This procedure will be repeated using the left wrist and the right side of the head.
Arm/Group | Botulinum Only | Botulinum Plus Physical Therapy
Number analyzed (Participants) | 8 | 8
units on a scale | 68 (16) | 88 (18)

3. Primary Outcome: Clinical Global Impression Scale (CGIS)
Description: This scale is an investigator-rated scale that measures illness severity on a single 7-point scale (1-7). Higher scores represent greater severity of illness.
Time Frame: absolute value at Week 12
Population: mean difference was calculated
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Only | Botulinum Plus Physical Therapy
Number analyzed (Participants) | 8 | 8
units on a scale | 3 (1) | 2 (1)

4. Secondary Outcome: Mean MEP After Paired Associative Stimulation (PASmean)
Description: A standard transcranial magnetic stimulation (TMS) paired associative stimulation (PAS) protocol was used to measure of neuroplasticity (the ability of the brain to form new connections). A nerve stimulator was placed on the wrist of the right hand to stimulate the median and ulnar nerves, set at the lowest intensity where the right thumb begins to twitch. An EMG sensor was placed over the abductor pollicis brevis muscle to measure muscle contractions. A magnetic coil was placed on the scalp on the left side of the head, overlying the brain's motor cortex, to stimulate the brain's output to the muscles in the opposite hand. 90 pairs of TMS and nerve stimulator pulses were applied. Then the motor evoked potential (MEP) from a single TMS pulse recorded from the surface EMG of the abductor pollicis brevis muscle was determined immediately, at 15 min and at 30 min after completion of the PAS protocol. The mean of these MEPs (PASmean) was compared between baseline and followup.
Time Frame: absolute value at week 12
Population: mean difference was calculated
Measure: Mean (Standard Deviation); unit: millivolts
Arm/Group | Botulinum Only | Botulinum Plus Physical Therapy
Number analyzed (Participants) | 8 | 8
millivolts | 1.7 (0.5) | 1.3 (0.6)

5. Other Pre Specified Outcome: Visual Analog Scale
Description: This is a single item scale, on which participants will mark the level of pain from 0-10. Higher score represents more severe pain.
Time Frame: absolute value at 12 weeks
Population: mean difference was calculated
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Only | Botulinum Plus Physical Therapy
Number analyzed (Participants) | 8 | 8
units on a scale | 6 (3) | 4 (2)

6. Other Pre Specified Outcome: Cervical Range of Motion Measurement
Description: Participants will be asked to sit in a chair and move the head to the left, to the right, to the front, and to the back. Then, participants be asked to tilt the head from side to side. A goniometer will be used to measure how far the head is able to move. The goniometer is similar to a protractor that measures magnitude of angle. A greater number indicates a greater range of motion. The minimum score would be 0, with no definite maximum (would not clinically be expected to exceed 70 degrees).
Time Frame: absolute value at 12 weeks was calculated
Population: mean difference was calculated
Measure: Mean (Standard Deviation); unit: Angle in degrees
Arm/Group | Botulinum Only | Botulinum Plus Physical Therapy
Number analyzed (Participants) | 8 | 8
Angle in degrees | 25 (14) | 26 (14)

ADVERSE EVENTS:
Arm/Group | Botox Only | Botox Plus Physical Therapy
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No